CLINICAL TRIAL: NCT00735787
Title: Controlled Study of Humira in Subjects With Chronic Plaque Psoriasis of the Hands and/or Feet
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Martin Okun MD, Director, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M10-405
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Results first posted 2010-11-01 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo/Adalimumab (Placebo Comparator): Loading dose of 2 placebo injections at Week 0 and placebo injections every other week (eow) from Week 1 through Week 15.
  In second period of study, subjects who continued in the study received 80 mg adalimumab at Week 16 followed by open-label 40 mg adalimumab eow from Week 17 to Week 27.
  Interventions: Biological: Placebo; Biological: Adalimumab
- Adalimumab (Active Comparator): 80 mg adalimumab loading dose at Week 0 and 40 mg adalimumab eow from Weeks 1 through 15. For subjects who continued in the second period of the study, subjects received 2 placebo injections at Week 16 to maintain the blind. Open-label 40 mg adalimumab eow was administered from Week 17 through Week 27.
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Placebo — Loading dose of 2 placebo subcutaneous (SC) injections (0.8 ml) at Week 0 followed by 1 injection SC eow from Week 1 to Week 15.In second period of study, subjects who continued in the study received 80 mg adalimumab at Week 16 followed by open-label 40 mg adalimumab eow from Week 17 to Week 27.
  Arms: Placebo/Adalimumab
Biological: Adalimumab — Loading dose of 80 mg adalimumab SC (two 40 mg injections) followed by 40 mg adalimumab SC eow.
  Other Names: Humira; ABT-D2E7

SUMMARY:
Evaluate the efficacy and safety of a 16-week course of Humira (adalimumab) compared to placebo in adults with chronic plaque psoriasis of the hands and/or feet and the sustainability of response for 12 additional weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult with Diagnosis of chronic plaque psoriasis of the Hands and Feet for at least 6 months, with a PGA >/=3 and candidates for systemic therapy;
* Patients in good general health
* Able to self-administer injections
* Negative chest x-ray (CXR) and purified protein derivative (PPD) test, unless willing to start anti-tuberculosis (TB) prophylaxis

Exclusion Criteria:

* Previous treatment with HUMIRA®
* Required mediation stability or washouts for: systemic corticosteroids (28 days), other investigational agent, other systemic therapies for psoriasis, ultraviolet B (UVB), psoralen with UVA (PUVA)
* Other active skin diseases or skin infections
* Diagnosis of palmoplantar pustulosis; erythrodermic psoriasis, pustular psoriasis, medication-induced or exacerbated psoriasis or new onset of guttate psoriasis
* Evidence of dysplasia or history of malignancy (Other than a successfully treated non-metastatic cutaneous squamous cell, basal cell carcinoma or localized carcinoma in situ of the cervix);
* History of listeriosis, histoplasmosis, chronic or active Hepatitis B infection, human immunodeficiency virus (HIV) infection, immunodeficiency syndrome, chronic recurring infections or active tuberculosis (TB);
* History of moderate to severe congestive heart failure,
* Recent cerebrovascular accident and any other condition which, in the opinion of the investigator, would put the subject at risk;
* History of central nervous system (CNS) demyelinating disease or neurologic symptoms suggestive of CNS demyelinating disease;
* History of clinically significant drug or alcohol abuse in the last 12 months;
* Infection(s) requiring treatment with intravenous (IV) antibiotics, IV antivirals, or IV antifungals within 30 days prior to Baseline or oral antibiotics, oral antivirals, or oral antifungals within 14 days prior to Baseline;
* Known hypersensitivity to the excipients of HUMIRA® as stated in the label;
* Female subjects who are pregnant or breast-feeding or considering becoming pregnant during the study.
* Prior exposure to Tysabri® (natalizumab)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Okun, MD, Study Director — Abbott
Locations (17):
- United States (8):
  - Site Reference ID/Investigator# 10168, Little Rock, Arkansas
  - Site Reference ID/Investigator# 10005, Bakersfield, California
  - Site Reference ID/Investigator# 10003, Macon, Georgia
  - Site Reference ID/Investigator# 10171, St Louis, Missouri
  - Site Reference ID/Investigator# 10164, East Windsor, New Jersey
  - Site Reference ID/Investigator# 10173, Dallas, Texas
  - Site Reference ID/Investigator# 11302, Houston, Texas
  - Site Reference ID/Investigator# 10166, San Antonio, Texas
- Canada (9):
  - Site Reference ID/Investigator# 10180, Edmonton, Alberta
  - Site Reference ID/Investigator# 10169, Vancouver, British Columbia
  - Site Reference ID/Investigator# 10170, Halifax, Nova Scotia
  - Site Reference ID/Investigator# 10179, Hamilton, Ontario
  - Site Reference ID/Investigator# 10004, London, Ontario
  - Site Reference ID/Investigator# 10177, North Bay, Ontario
  - Site Reference ID/Investigator# 10175, Waterloo, Ontario
  - Site Reference ID/Investigator# 10165, Montreal, Quebec
  - Site Reference ID/Investigator# 10176, Québec, Quebec

REFERENCES:
- [Derived] Leonardi C, Langley RG, Papp K, Tyring SK, Wasel N, Vender R, Unnebrink K, Gupta SR, Valdecantos WC, Bagel J. Adalimumab for treatment of moderate to severe chronic plaque psoriasis of the hands and feet: efficacy and safety results from REACH, a randomized, placebo-controlled, double-blind trial. Arch Dermatol. 2011 Apr;147(4):429-36. doi: 10.1001/archdermatol.2010.384. Epub 2010 Dec 20. PMID 21173304
- See also: prescribing information — http://www.humira.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Adalimumab: Placebo injections every other week (eow) up to Week 15. In second period of study, subjects who continued to participate received 80 mg adalimumab at Week 16 followed by open-label 40 mg adalimumab eow from Week 17 to Week 27.
- Adalimumab: 80 mg adalimumab loading dose at Week 0 and 40 mg adalimumab eow from Weeks 1 through 27. Subjects received 2 placebo injections at Week 16 to maintain the blind.
Period: Period 1
Arm/Group | Placebo/Adalimumab | Adalimumab
Started | 23 | 49
Completed | 17 (Per visit window, 18 completed; 17 completed per subject case report form.) | 41
Not Completed | 6 | 8
Period: Period 2
Arm/Group | Placebo/Adalimumab | Adalimumab
Started | 18 | 41
Completed | 13 | 40
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Adalimumab | Adalimumab | Total
Number analyzed (Participants) | 23 | 49 | 72
Age Categorical [Number; unit: subjects]
  < 40 years | 1 | 11 | 12
  Between 40 and < 60 years | 14 | 29 | 43
  >= 60 years | 8 | 9 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 54.8 (11.40) | 49.0 (11.41) | 50.9 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 28 | 43
  Male | 8 | 21 | 29
Region of Enrollment [Number; unit: participants]
  United States | 9 | 20 | 29
  Canada | 14 | 29 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Physician's Global Assessment of Psoriasis (PGA) of Clear or Almost Clear at Week 16
Description: Number of subjects achieving a PGA of clear (representing no signs of plaque psoriasis) or almost clear (representing just perceptible erythema and scaling) at Week 16. The PGA is a 5-point scale used to measure the severity of disease at the time of the physician's evaluation of the subject. The degree of overall severity is rated as follows: 0-Clear, 1-Almost clear, 2-Mild, 3-Moderate, and 4-Severe.
Time Frame: Week 16
Population: Analysis was based on the intention to treat (ITT) subject population. Subjects who did not achieve PGA assessments at Week 16 were imputed as non-responders.
Measure: Number; unit: subjects
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
subjects | 1 | 15
Statistical Analysis 1: Comparison: Placebo/Adalimumab vs Adalimumab; The primary null hypothesis for this study was that there was no difference in the proportion of subjects that achieved PGA clear or almost clear at Week 16 between the adalimumab and placebo groups. Analysis was done using a two-sided Fisher's exact test at alpha level=0.05; Test type: Superiority or Other; p = 0.014, Fisher Exact

2. Secondary Outcome: Mean Change From Baseline in Erythema, Scaling, Induration, and Fissuring (ESIF)
Description: Severity of each sign of ESIF was assessed using a 4-point scale (0 = clear, 1 = mild, 2 = moderate, and 3 = severe). The ESIF was calculated by adding the scores for the 4 signs for the two soles and two palms, for a total range from 0 (no disease) to 48 points (most severe condition). A decrease from Baseline in ESIF indicates improvement.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 28
Population: Analysis was based on the ITT subject population and performed using last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
units on a scale
  Week 2 | -2.35 (4.074) | -6.24 (7.685)
  Week 4 | -1.91 (7.019) | -7.73 (9.064)
  Week 8 | -3.04 (7.327) | -9.33 (9.335)
  Week 12 | -5.30 (6.825) | -10.80 (11.175)
  Week 16 | -5.04 (6.568) | -10.92 (12.460)
  Week 20 (open-label) | -6.43 (8.805) | -11.69 (11.353)
  Week 24 (open-label) | -5.83 (9.267) | -11.51 (11.502)
  Week 28 (open-label) | -5.83 (8.574) | -11.96 (10.261)

3. Secondary Outcome: Mean Change From Baseline in ESIF for Palms
Description: Severity of each sign of ESIF was assessed using a 4-point scale (0 = clear, 1 = mild, 2 = moderate, and 3 = severe). The ESIF was calculated by adding the scores for the 4 signs for the palms of the hands, yielding a total range from 0 (no disease) to 24 points (most severe condition) for the palms. A decrease from Baseline in ESIF indicates improvement.
Time Frame: Baseline and Weeks 2, 4, 12, 16, 20, 24, and 28
Population: Analysis was based on the ITT subject population and performed using the LOCF method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
units on a scale
  Week 2 | -1.78 (3.464) | -3.33 (4.095)
  Week 4 | -1.57 (4.326) | -4.33 (4.543)
  Week 8 | -2.09 (4.889) | -5.35 (4.829)
  Week 12 | -3.39 (4.639) | -5.53 (5.934)
  Week 16 | -2.65 (4.914) | -5.80 (6.285)
  Week 20 (open-label) | -3.87 (5.810) | -6.16 (5.669)
  Week 24 (open-label) | -3.74 (5.387) | -6.08 (5.947)
  Week 28 (open-label) | -3.52 (4.870) | -6.59 (5.244)

4. Secondary Outcome: Mean Change From Baseline in ESIF for Soles
Description: Severity of each sign of ESIF was assessed using a 4-point scale (0 = clear, 1 = mild, 2 = moderate, and 3 = severe). The ESIF was calculated by adding the scores for the 4 signs for the soles of the feet, yielding a total range from 0 (no disease) to 24 points (most severe condition) for the soles. A decrease from Baseline in ESIF indicates improvement.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 28
Population: Analysis was based on the ITT subject population and performed using the LOCF method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
units on a scale
  Week 2 | -0.57 (1.619) | -2.92 (4.650)
  Week 4 | -0.35 (3.915) | -3.39 (5.553)
  Week 8 | -0.96 (4.017) | -4.04 (5.972)
  Week 12 | -1.91 (3.965) | -5.35 (6.515)
  Week 16 | -2.39 (4.620) | -5.18 (7.132)
  Week 20 (open-label) | -2.57 (5.358) | -5.47 (6.959)
  Week 24 (open-label) | -2.09 (5.608) | -5.37 (7.082)
  Week 28 (open-label) | -2.30 (5.431) | -5.31 (6.378)

5. Secondary Outcome: Number of Subjects With Moderate Improvement in ESIF From Baseline
Description: Number of subjects that achieved > 50% reduction from Baseline in ESIF.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 28
Population: Analysis was based on the ITT subject population and performed using non-responder imputation (NRI).
Measure: Number; unit: subjects
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
subjects
  Week 2 | 1 | 8
  Week 4 | 2 | 10
  Week 8 | 3 | 17
  Week 12 | 6 | 20
  Week 16 | 4 | 21
  Week 20 (open-label) | 6 | 19
  Week 24 (open-label) | 6 | 21
  Week 28 (open-label) | 3 | 19

6. Secondary Outcome: Number of Subjects With Marked Improvement in ESIF From Baseline
Description: Number of subjects that achieved > 75% reduction from Baseline in ESIF
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 28
Population: Analysis was based on the ITT subject population and performed using non-responder imputation (NRI).
Measure: Number; unit: subjects
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
subjects
  Week 2 | 0 | 3
  Week 4 | 0 | 5
  Week 8 | 0 | 7
  Week 12 | 0 | 11
  Week 16 | 1 | 14
  Week 20 (open-label) | 5 | 13
  Week 24 (open-label) | 4 | 12
  Week 28 (open-label) | 2 | 11

7. Secondary Outcome: Mean Change From Baseline in Nail Psoriasis Severity Index (NAPSI)
Description: For subjects with psoriasis nail involvement at Baseline, the target fingernail (most severely involved fingernail at Baseline) was assessed for NAPSI throughout the study. NAPSI ranges from 0 (no nail psoriasis) to 8 (most severe nail psoriasis).
Time Frame: Baseline and Weeks 8, 16, and 28
Population: Analysis was performed in the ITT subject population for subjects with nail involvement at baseline only and is based on LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 8 | 28
units on a scale
  Week 8 | -0.63 (1.061) | -0.88 (1.211)
  Week 16 | -0.13 (1.246) | -1.67 (1.593)
  Week 28 (open-label) | -1.00 (1.852) | -2.00 (2.177)

8. Secondary Outcome: Number of Subjects With Physicians Global Assessment of Psoriasis (PGA) of Clear, Almost Clear, or Mild
Description: Number of subjects achieving a PGA of clear (representing no signs of plaque psoriasis), almost clear (representing just perceptible erythema and scaling), or mild (representing light pink erythema with minimal scaling and with or without pustules). The PGA is a 5-point scale used to measure the severity of disease at the time of the physician's evaluation of the subject. The degree of overall severity is rated as follows: 0-Clear, 1-Almost clear, 2-Mild, 3-Moderate, and 4-Severe.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, and 28
Population: Analysis was based on the ITT subject population and performed using non-responder imputation (NRI).
Measure: Number; unit: subjects
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
subjects
  Week 2 | 2 | 15
  Week 4 | 3 | 21
  Week 8 | 6 | 21
  Week 12 | 8 | 24
  Week 16 | 6 | 25
  Week 20 (open-label) | 8 | 23
  Week 24 (open-label) | 7 | 20
  Week 28 (open-label) | 4 | 23

9. Secondary Outcome: Number of Subjects With PGA of Clear or Almost Clear
Description: Number of subjects achieving a PGA of clear (representing no signs of plaque psoriasis) or almost clear (representing just perceptible erythema and scaling). The PGA is a 5-point scale used to measure the severity of disease at the time of the physician's evaluation of the subject. The degree of overall severity is rated as follows: 0-Clear, 1-Almost clear, 2-Mild, 3-Moderate, and 4-Severe.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 20, 24, and 28
Population: Analysis was based on the ITT subject population and performed using non-responder imputation (NRI).
Measure: Number; unit: subjects
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
subjects
  Week 2 | 1 | 4
  Week 4 | 1 | 10
  Week 8 | 2 | 12
  Week 12 | 3 | 14
  Week 20 (open-label) | 5 | 11
  Week 24 (open-label) | 5 | 12
  Week 28 (open-label) | 2 | 12

10. Secondary Outcome: Number of Subjects With PGA of Clear
Description: Number of subjects achieving a PGA of clear (representing no signs of plaque psoriasis). The PGA is a 5-point scale used to measure the severity of disease at the time of the physician's evaluation of the subject. The degree of overall severity is rated as follows: 0-Clear, 1-Almost clear, 2-Mild, 3-Moderate, and 4-Severe.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, and 28
Population: Analysis was based on the ITT subject population and performed using NRI.
Measure: Number; unit: subjects
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
subjects
  Week 2 | 0 | 1
  Week 4 | 0 | 2
  Week 8 | 0 | 3
  Week 12 | 0 | 6
  Week 16 | 1 | 6
  Week 20 (open-label) | 2 | 8
  Week 24 (open-label) | 3 | 7
  Week 28 (open-label) | 2 | 7

11. Secondary Outcome: Number of Subjects With Psoriasis Area and Severity Index (PASI) 50
Description: Number of subjects who achieved 50% or greater improvement from baseline PASI. The PASI scale is from 0 (no psoriasis) to 72 (complete erythroderma of the severest possible degree).
Time Frame: Baseline and Weeks 16 and 28
Population: Analysis was based on the ITT subject population and performed using NRI.
Measure: Number; unit: subjects
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
subjects
  Week 16 | 5 | 21
  Week 28 (open-label) | 8 | 21

12. Secondary Outcome: Number of Subjects With PASI 75
Description: Number of subjects who achieved 75% or greater improvement from baseline PASI. The PASI scale is from 0 (no psoriasis) to 72 (complete erythroderma of the severest possible degree).
Time Frame: Baseline and Weeks 16 and 28
Population: Analysis was based on the ITT subject population and performed using NRI.
Measure: Number; unit: subjects
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
subjects
  Week 16 | 2 | 15
  Week 28 (open-label) | 4 | 11

13. Secondary Outcome: Number of Subjects With PASI 90
Description: Number of subjects who achieved 90% or greater improvement from baseline PASI. The PASI scale is from 0 (no psoriasis) to 72 (complete erythroderma of the severest possible degree).
Time Frame: Baseline and Weeks 16 and 28
Population: Analysis was based on the ITT subject population and performed using NRI.
Measure: Number; unit: subjects
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
subjects
  Week 16 | 0 | 10
  Week 28 (open-label) | 4 | 10

14. Secondary Outcome: Number of Subjects With PASI 100
Description: Number of subjects who achieved 100% improvement from baseline PASI. The PASI scale is from 0 (no psoriasis) to 72 (complete erythroderma of the severest possible degree).
Time Frame: Baseline and Weeks 16 and 28
Population: Analysis was based on the ITT subject population and performed using NRI.
Measure: Number; unit: subjects
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
subjects
  Week 16 | 0 | 7
  Week 28 (open-label) | 1 | 8

15. Secondary Outcome: Mean Change From Baseline in Dermatology Life Quality Index (DLQI)
Description: The DLQI consists of 10 questions and is scored from 0 (total lack of impairment) to 30 (life is very much impaired). A decrease in DLQI indicates improvement.
Time Frame: Baseline and Weeks 2, 8, 16, and 28
Population: Analysis was based on the ITT subject population and performed using LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
units on a scale
  Week 2 | -3.43 (3.435) | -4.35 (4.741)
  Week 8 | -3.09 (5.008) | -4.08 (5.541)
  Week 16 | -4.22 (4.936) | -4.78 (7.269)
  Week 28 (open-label) | -4.74 (4.731) | -5.18 (7.499)

16. Secondary Outcome: Number of Subjects Achieving a DLQI of 0
Description: Number of subjects achieving a DLQI score of 0, indicating total lack of impairment. The DLQI consists of 10 questions and is scored from 0 to 30 (life is very much impaired). A decrease in DLQI indicates improvement.
Time Frame: Baseline and Weeks 2, 8, 16, and 28
Population: Analysis was based on the ITT subject population and performed using NRI.
Measure: Number; unit: subjects
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
subjects
  Week 2 | 1 | 3
  Week 8 | 1 | 3
  Week 16 | 0 | 7
  Week 28 (open-label) | 1 | 6

17. Secondary Outcome: Mean Change From Baseline in Visual Analog Scale (VAS) for Psoriasis and Psoriatic Arthritis Pain
Description: On one single VAS, subjects assessed their pain due to psoriasis (and psoriatic arthritis, if applicable). Mean change in psoriasis and psoriatic arthritis pain from Baseline as measured by a VAS from 0 (no pain) to 100 (pain as bad as it could be).
Time Frame: Baseline and Weeks 16 and 28
Population: Analysis was based on the ITT subject population and performed using LOCF.
Measure: Mean (Standard Deviation); unit: mm on scale
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
mm on scale
  Week 16 | -12.45 (28.637) | -17.49 (34.451)
  Week 28 (open-label) | -16.25 (24.950) | -16.59 (34.430)

18. Secondary Outcome: Mean Change From Baseline in Work Productivity and Activity Impairment Questionnaire: Psoriasis (WPAI:PSO)
Description: WPAI:PSO assesses the effect on the subject's ability to work and perform regular activities in 4 areas: % work time (in hours) missed due to psoriasis, % impairment while working (on a scale from 0 [psoriasis having no effect] to 10 [psoriasis completely prevented subject from working]), % overall work impairment (on a scale from 0 [psoriasis having no effect] to 10 [psoriasis completely prevented subject from working]), and % activity impairment (on a scale from 0 [psoriasis having no effect on daily activities] to 10 [psoriasis completely prevented subject from doing daily activities]).
Time Frame: Baseline and Weeks 8, 16, and 28
Population: Analysis was based on the ITT subject population and performed using LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
units on a scale
  % Work Time Missed due to Psoriasis Week 8 | 6.32 (24.953) | 4.70 (12.778)
  % Work Time Missed due to Psoriasis Week 16 | 7.72 (33.299) | 5.34 (20.250)
  % Work Time Missed due to Psoriasis Week 28 (OL) | 2.60 (26.628) | 3.16 (18.198)
  % Impairment While Working Week 8 | 0.71 (29.733) | -8.21 (27.087)
  % Impairment While Working Week 16 | -4.67 (20.656) | -5.94 (27.103)
  % Impairment While Working Week 28 (OL) | -5.33 (20.999) | -8.44 (31.429)
  % Overall Work Impairment Week 8 | -0.48 (29.988) | -8.97 (27.355)
  % Overall Work Impairment Week 16 | -5.45 (22.432) | -7.19 (26.556)
  % Overall Work Impairment Week 28 (OL) | -5.79 (20.996) | -9.88 (31.045)
  % Activity Impairment Week 8 | -9.09 (32.500) | -11.02 (23.562)
  % Activity Impairment Week 16 | -9.09 (22.234) | -13.88 (27.600)
  % Activity Impairment Week 28 (OL) | -15.91 (27.196) | -14.69 (32.539)

19. Secondary Outcome: Mean Change From Baseline in Patient Health Questionnaire (PHQ-9)
Description: The PHQ-9 consists of 9 questions that assess how often over the past 2 weeks subjects had signs or symptoms of depression (0=not at all, 1=several days, 2=more than half days, and 3=nearly every day). The PHQ-9 is the sum of the scores from the 9 questions for a total range from 0 (not depressed at all) to 27 (depressed nearly every day).
Time Frame: Baseline and Weeks 2, 8, 16, and 28
Population: Analysis was based on the ITT subject population and performed using LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
units on a scale
  Week 2 | -2.85 (4.332) | -2.86 (4.449)
  Week 8 | -2.43 (4.057) | -1.80 (4.796)
  Week 16 | -2.64 (6.637) | -2.14 (4.659)
  Week 28 (open-label) | -3.32 (5.719) | -2.65 (5.031)

20. Secondary Outcome: Number of Subjects With Difficulties According to PHQ-9
Description: Based on the 9 questions of the PHQ-9, if subjects indicated any problems (PHQ-9 score > 0), the difficulty to do work, take care of things at home, and get along with people (question 10 of the PHQ) were assessed (not difficult at all, somewhat difficult, very difficult, and extremely difficult).
Time Frame: Baseline and Weeks 2, 8, 16, and 28
Population: Analysis was based on the ITT subject population. Missing values were imputed as "extremely difficult."
Measure: Number; unit: subjects
Arm/Group | Placebo/Adalimumab | Adalimumab
Number analyzed (Participants) | 23 | 49
subjects
  Not difficult at all - Baseline | 4 | 20
  Somewhat difficult - Baseline | 9 | 19
  Very difficult - Baseline | 3 | 5
  Extremely difficult - Baseline | 7 | 5
  Not difficult at all - Week 2 | 5 | 21
  Somewhat difficult - Week 2 | 9 | 16
  Very difficult - Week 2 | 2 | 3
  Extremely difficult - Week 2 | 7 | 9
  Not difficult at all - Week 8 | 4 | 18
  Somewhat difficult - Week 8 | 8 | 15
  Very difficult - Week 8 | 2 | 5
  Extremely difficult - Week 8 | 9 | 11
  Not difficult at all - Week 16 | 3 | 19
  Somewhat difficult - Week 16 | 8 | 10
  Very difficult - Week 16 | 2 | 1
  Extremely difficult - Week 16 | 10 | 19
  Not difficult at all - Week 28 (OL) | 4 | 21
  Somewhat difficult - Week 28 (OL) | 5 | 6
  Very difficult - Week 28 (OL) | 2 | 1
  Extremely difficult - Week 28 (OL) | 12 | 21

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) from the time of study drug administration until 70 days following completion (Week 28) or discontinuation of study drug administration.
Description: For subjects who continued adalimumab therapy (commercial) after discontinuation of study treatment, AEs that occurred after the first dose of non-study provided adalimumab were not to be report in this study, but rather via the usual post-marketing reporting process.
Arm/Group | Placebo/Adalimumab | Adalimumab
Serious Adverse Events (participants affected / at risk) | 1/23 | 2/49
Other Adverse Events (participants affected / at risk) | 15/23 | 30/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Adalimumab (N=23) | Adalimumab (N=49)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Adalimumab (N=23) | Adalimumab (N=49)
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Toothache (Gastrointestinal disorders) | 2 | 0
Injection site reaction (General disorders) | 2 | 2
Oedema peripheral (General disorders) | 2 | 2
Bronchitis (Infections and infestations) | 3 | 1
Gastroenteritis (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 3 | 13
Pharyngitis (Infections and infestations) | 1 | 3
Sinusitis (Infections and infestations) | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 2 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Headache (Nervous system disorders) | 1 | 7
Insomnia (Psychiatric disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 3

LIMITATIONS AND CAVEATS:
Based on one investigator's non-compliance with the protocol at one site, ITT analyses were conducted in a smaller number of subjects that excluded all 9 subjects from this one site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.